CLINICAL TRIAL: NCT05027451
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Single-Dose Intravenous Study to Evaluate the Safety and Pharmacokinetics of IXT-m200 in Healthy Participants
Brief Title: Safety, Tolerability, and Pharmacokinetics of IXT-m200
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InterveXion Therapeutics, LLC (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: M200C-2102; U01DA045366 (NIH)
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IXT-m200 (Experimental): 3 g of IXT-m200 given once by 30-min intravenous infusion
  Interventions: Drug: IXT-m200
- Placebo (Placebo Comparator): Normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: IXT-m200 — Anti-methamphetamine chimeric monoclonal antibody (mAb)
  Other Names: ch-mAb7F9
  Arms: IXT-m200
Other: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
Approximately 9 participants will be enrolled in the study in a single cohort. Participants will be randomized to 3 g IXT-m200 or placebo at 7:2. Each will receive their dose as a 30-min intravenous infusion, then remain at the study site overnight to complete Day 1 and Day 2 assessments (e.g., electrocardiogram (ECG), laboratory assessments, blood draws, and vital signs). Following discharge on Day 2, participants will return to the clinic for follow-up pharmacokinetic (PK) and safety assessments on Day 8, then every 1-3 weeks thereafter until Day 127.

ELIGIBILITY:
Inclusion Criteria:

-

Eligible participants will:

1. Be 18-65 years of age, inclusive, at the time of study consent;
2. Be able and willing to read, comprehend, and give Authorization for Use/Disclosure of Health Information (HIPAA) and informed consent;
3. Be healthy, based on the pre-study medical evaluation (medical history and physical exam, vital signs, ECG, and clinical laboratory evaluations);
4. Be willing to comply with study instructions and dosing, agree to make all appointments, and complete the entire course of the study;
5. Be of nonchildbearing potential or agree to use protocol-specified method(s) of birth control throughout study participation;
6. Agree to adhere to Lifestyle Considerations throughout study duration.

Exclusion Criteria:

-

Eligible participants will NOT:

1. Have a history of treatment with a monoclonal antibody in the past year;
2. Have a known contraindication or sensitivity to IXT-m200 based on known allergies to other mAbs, any inactive ingredient of IXT-m200, or any other products required for the study procedures;
3. Have a history of alcohol and/or drug use disorder, as determined by DSM-5 criteria;
4. Have a history of stimulant use, including methamphetamine and amphetamine;
5. Be currently taking certain other drugs and medications, including: "designer drugs" (e.g., 3,4-methylenedioxyMETH (MDMA, Ecstasy, Adam, XTC) and its N-dimethyl metabolite methylenedioxyamphetamine (MDA), anti-orexigenic drugs (including over-the-counter medications for weight loss), or be chronic users of phenethylamine compounds (e.g., phenylpropanolamine, ephedrine, pseudoephedrine, amphetamine, phentermine, phenmetrazine, methylphenidate, diethylpropion, and propylhexedrine);
6. Have a positive drug screen for any psychoactive substances (legal or nonlegal) on Day 1 prior to dosing;
7. Have a history of severe allergy (rash, hives, breathing difficulty, etc) to any medications;
8. Have a history of allergic or environmental bronchial asthma within the past 3 years;
9. Have a clinically significant history of or current abnormality or disease of any organ system, including renal, hepatic, gastrointestinal, cardiovascular, pulmonary (including chronic asthma), endocrine (eg, diabetes), central nervous (eg psychiatric conditions), or hematologic systems, or recent clinically significant surgery;
10. Have a history of seizure, epilepsy, severe head injury, multiple sclerosis, or other known neurological conditions;
11. Have a planned or scheduled surgical procedure during the study;
12. Have recently donated blood or plasma (within 30 days of study drug dose);
13. Have a current diagnosis of anorexia nervosa or bulimia disorder;
14. Be currently participating or has participated within the last 30 days prior to the start of this study in a drug, device, or other interventional research study;
15. Be pregnant or lactating;
16. In the Investigator's or Sponsor's (or designee) opinion, be inappropriate for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — InterveXion Therapeutics
Locations (1):
- Clinilabs Drug Development Corporation, Eatontown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Final datasets are expected to contain pharmacokinetic data on IXT-m200 and safety data. No individually identifiable private information will be distributed.
Time Frame: These datasets will be available for distribution following submission to the FDA of the Clinical Study Report and publication. They will be available for 2 years after the initial publication.
Access Criteria: These datasets and associated documentation will be made available on CD by the Sponsor to requestors under a data sharing agreement that provides for: (1) a commitment to using the data only for research purposes; (2) a commitment to securing the data using appropriate computer technology and not distributing to third parties; and (3) a commitment to destroying or returning the data after analyses are completed. Requests should be sent to intervexion@gmail.com.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants underwent screening procedures to check eligibility criteria within 30 days prior to randomization.
Period: Overall Study
Arm/Group | IXT-m200 | Placebo
Started | 7 | 2
Completed | 6 | 1
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline assessments were conducted at the screening visit or on Day 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | IXT-m200 | Placebo | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (8.75) | 42.5 (13.44) | 42.0 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 5
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 2 | 1 | 3
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 2 | 9
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.7 (2.67) | 24.38 (4.91) | 28.52 (3.72)
Weight [Mean (Standard Deviation); unit: kg] | 87.41 (9.83) | 64 (4.1) | 82.21 (13.46)
Height [Mean (Standard Deviation); unit: cm] | 171.5 (5.91) | 163 (11.31) | 169.59 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events (AEs) Assessed by Physical Examinations
Description: Physical examinations
Time Frame: 127 days
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | IXT-m200 | Placebo
Number analyzed (Participants) | 7 | 2
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-related AEs Assessed by Vital Signs
Description: Blood pressure, heart rate, and temperature
Time Frame: 127 days
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | IXT-m200 | Placebo
Number analyzed (Participants) | 7 | 2
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Treatment-related AEs Assessed by ECG
Description: Electrocardiogram
Time Frame: 30 min post-dose completion
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | IXT-m200 | Placebo
Number analyzed (Participants) | 7 | 2
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Treatment-related AEs Assessed by Clinical Laboratory Testing
Description: Clinical laboratory testing
Time Frame: 64 days
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | IXT-m200 | Placebo
Number analyzed (Participants) | 7 | 2
Participants | 1 | 0

5. Secondary Outcome: Time Course of IXT-m200 Concentrations
Description: IXT-m200 concentrations over time
Time Frame: 127 days
Population: All participants receiving IXT-m200
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | IXT-m200
Number analyzed (Participants) | 7
mg/L
  Pre-dose | 0 (0)
  1 hr post-dose | 728 (157)
  4 hr post-dose | 705 (100)
  8 hr post-dose | 632 (104)
  Day 2 | 632 (132)
  Day 8 | 316 (62.6)
  Day 15 | 257 (31)
  Day 22 | 194 (48)
  Day 29 | 155 (50.9)
  Day 36 | 109 (22.5)
  Day 43 | 84.1 (14.8)
  Day 64: number analyzed (Participants) | 5
  Day 64 | 37.4 (12.2)
  Day 85 | 13.5 (4.3)
  Day 106 | 6.92 (1.98)
  Day 127: number analyzed (Participants) | 6
  Day 127 | 3.65 (1.4)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected following the start of administration of study drug on Day 1 through the final study visit on Day 127.
Description: AE data were collected at study visits or between visits if participants informed the site by phone or visit.
Arm/Group | IXT-m200 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/2
Other Adverse Events (participants affected / at risk) | 4/7 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IXT-m200 (N=7) | Placebo (N=2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SARS-CoV-2 antibody test positive (Investigations) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may prepare and submit manuscripts or slide shows based on Study Data. Such manuscripts or slide shows shall be submitted to Sponsor for review, at which time these may be approved or rejected. PI will not release those that are rejected by Sponsor. One investigator may be identified as an author or co-author of Sponsor-sponsored publications resulting from this study.

DOCUMENTS (3):
  • Study Protocol (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT05027451/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT05027451/SAP_001.pdf
  • Informed Consent Form (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT05027451/ICF_002.pdf